CLINICAL TRIAL: NCT03855293
Title: Protecting the Corneal Endothelium During Cataract Surgery Using the Anterior Capsule: a Prospective Randomised Double-masked Study
Brief Title: Protecting the Corneal Endothelium During Cataract Surgery Using the Anterior Capsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr., Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rhexis Protection Shield
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Endothelial Cell Loss, Corneal
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Other): rhexis protection shield
  Interventions: Procedure: Rhexis protection shield
- Control group (No Intervention): regular surgery

INTERVENTIONS:
Procedure: Rhexis protection shield — In the study group the anterior capsule will be used as a protection shield during pacoemulsifikation and removed after the phacoemulsifikation
  Arms: Study group

SUMMARY:
Cataract surgery is one of the most frequently performed surgical procedures worldwide. Since the introduction of phacoemulsification to remove the cataractous lens, risk and complication rates of cataract surgery decreased significantly.

The phacoemulsification technique utilizes a high-intensity ultrasound energy for the fragmentation and emulsification of the lens. One of the main complications during phacoemulsification, is damaging of the endothelium due to contact with lens fragments of the nucleus following turbulent flow of irrigating solution, resulting in corneal damage, inflammation of the endothelium and corneal edema.

In this study we want to evaluate the effect of the anterior capsule, gained by capsular rhexis, as a corneal shield during phacoemulsification on the corneal endothelium.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Written informed consent prior to surgery
* Moderate to severe nuclear or mixed cataract

Exclusion Criteria:

* Corneal pathologies
* Pregnancy
* Patients with an increased surgical risk (i.e. patients with pseudoexfoliation syndrome, patients with the potential risk of intra-operative floppy iris syndrome)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
endothelium cell loss | 1 year
  Comparison of the lost endothelium cells in both groups

SECONDARY OUTCOMES:
central corneal thickness | 1 year
  Comparison of corneal thickness between both groups